CLINICAL TRIAL: NCT03349242
Title: Natural History Study of Patients With X-linked Retinal Dystrophy Associated With Mutations in Retinitis Pigmentosa GTPase Regulator (RPGR)
Status: Completed | Type: Observational
Sponsor: MeiraGTx UK II Ltd (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: MGT011
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rod-cone dystrophies (often referred to as retinitis pigmentosa (RP)) are a clinically and genetically heterogeneous group of disorders in which there is progressive loss of rod and later cone photoreceptor function leading to severe visual impairment. RP usually occurs as an isolated retinal disorder, but it may also be seen in association with systemic abnormalities.

DETAILED DESCRIPTION:
X-linked Retinitis Pigmentosa (XLRP) is a severe form of RP with early onset of nyctalopia and progression to legal blindness by the 3rd to 4th decade. Most affected males show symptomatic night blindness before the age of 10 years, are often myopic and show fundus abnormalities and ERG changes in early childhood. Examination of close female relatives is helpful in the absence of a family history, as the recognition of the XL carrier state will confirm the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females aged 5 years or older
* Have RPGR-associated retinal dystrophy
* Are able to give informed consent or assent, with the guidance of their parent/guardian where appropriate
* Are able to undertake age-appropriate clinical assessments as specified in the protocol
* Have genetic mutation within the RPGR gene confirmed by an accredited lab or research lab.

Exclusion Criteria:

* Are unable or unwilling to undertake consent or clinical testing

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RPGR-associated retinal dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Analysis of retinal structure and function to assess disease progression | 6 years
  Retinal structure will be measured using Adaptive optics and SD-OCT and Fundal autofluorescence.

SECONDARY OUTCOMES:
Retinal Sensitivity | 6 years
  To be assessed by Microperimetry
Retinal Structural detailed phenotyping | 6 years
  Retinal Structure measured by Adaptive Optics (
Fundus Autofluorescence | 6 years
  Presence or Absence
Visual Fields testing | 6 years
  Assessment of Visual Fields with analysis of hill vision by perimetry

CONTACTS AND LOCATIONS:
Overall Officials: Michel Michaelides, Prof, Principal Investigator — UCL/Moorfields
Locations (8):
- United States (6):
  - Shiley Eye Institute - UCSD, La Jolla, California
  - Stanford University, Spencer Center for Vision Research, Stanford, California
  - Emory Eye Centre, Atlanta, Georgia
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Kellogg Eye Center, Ann Arbor, Michigan
  - UPMC Eye Centre, Pittsburgh, Pennsylvania
- The Hospital for Sick Children, Toronto, Canada
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided